CLINICAL TRIAL: NCT01715883
Title: Sodium Nitrite Administration at the Time of Lung Organ Procurement and Transplantation to Minimize the Risk of Pulmonary Graft Dysfunction
Brief Title: Sodium Nitrite in Lung Transplant Patients to Minimize the Risk of Pulmonary Graft Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of support staff
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Matthew Morrell, Assistant Professor, Department of Medicine, Division of Pulmonary, Allergy and Critical care medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO11030251
Record Dates: First submitted 2012-10-08; First posted 2012-10-29 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-05

CONDITIONS: Primary Graft Dysfunction
Keywords: Lung transplant; Pulmonary Graft Dysfunction; Sodium Nitrite
MeSH Terms: conditions — Primary Graft Dysfunction | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Nitrite (Experimental): Sodium Nitrite will be administered at three time points:
  At the time of organ procurement, a pre-prepared syringe of sodium nitrite will be added to each of the 2.8 liter bags of Perfadex solution to flush the donor lungs.
  At the time of transplant just prior to reperfusion of lungs, the donor lungs are flushed with a cold pneumoplegia solution after the bronchial (1st) anastomosis and with warm pneumoplegia solution after the portal vein (3rd, last) anastomosis. The drug will be added to pneumoplegia solution just prior to both the flushes.
  Sodium Nitrite will be delivered intravenously to the recipient immediately prior to lung reperfusion as a single infusion at rate of 4 mL/min for the first 30 min, followed by 2.2 mL/min for the next 60 min.
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite — Same as the details in Arm Description.

SUMMARY:
This is a Phase 2 observational nonrandomized pilot investigation to evaluate the safety and efficacy of Sodium Nitrite administration for the reduction of Primary Graft Dysfunction (PGD) in patients undergoing lung transplant. The study will enroll 8 subjects, undergoing lung transplant at the University of Pittsburgh Medical Center (UPMC).

DETAILED DESCRIPTION:
While increasing numbers of patients with advanced lung disease are candidates for lung transplantation, the short- and long-term outcomes are severely compromised by graft dysfunction, primarily in the form of organ rejection. The earliest manifestation of lung allograft dysfunction, termed primary graft dysfunction (PGD), represents a form of ischemia-reperfusion acute lung injury, and occurs in its severest form (Grade 3) in from 10 to 35% of lung transplant recipients 1-6. PGD is the primary cause of early morbidity and mortality after transplantation and is strongly associated with the late development of chronic lung rejection or Bronchiolitis Obliterans Syndrome (BOS. Early graft dysfunction contributes significantly to the suboptimal outcomes of lung transplantation and to the failure of lung transplant recipients to achieve five-year survival rates comparable to patients who receive other solid organs such as the heart and liver. The risk of PGD further limits the time that lungs can be stored ex-vivo, therefore restricting the pool of available donors. A critical advance in the prevention of both early and late lung allograft dysfunction will occur if PGD can be successfully prevented or minimized.

In this study, the investigators propose to test the hypothesis that administration of Sodium Nitrite to donor lungs and lung transplant recipients at the time of transplantation will be safe and will reduce the incidence of grades 2 and 3 PGD, thereby improving clinical outcomes with minimal toxicity.

Sodium Nitrite will be obtained from a commercial preparation (Hope Pharmaceuticals) and the UPMC Pharmacy will prepare the formulations, which will be infused at three time points. First it will be infused into the preservation solution bag at the time of organ procurement from the donor, then to the allograft at the time of transplantation, and finally as a direct infusion into the organ recipient.

The investigators plan to enroll total of 8 subjects undergoing lung transplantation for this Phase 2 observational non-randomized pilot investigation to evaluate the safety, efficacy, and pharmacokinetics of Sodium Nitrite administration when administered to the procured lung and lung transplant recipient, for the prevention of Primary Graft Dysfunction (PGD). It is anticipated that positive results from this trial lead to a larger clinical investigation of Sodium Nitrite administration directed at producing a reduction in PGD and perhaps secondary obliterative bronchiolitis; and will potentially allow for extended organ storage, extended use of more marginal organs, and more effective use of Donation after Cardiac Death (DCD) organs which undergo combination of warm and cold ischemia for organ procurement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing lung transplantation.
* Subjects in the age range of 18-70 years
* Ability to understand and provide consent. Proxy consent will not be accepted.

Exclusion Criteria:

* Donor exclusion criteria
* Age > 55 years.
* Mechanical ventilation > 5 days prior to procurement
* Significant chest trauma or lung contusion
* Smoking history > 20 pack-year
* Ratio of arterial oxygen partial pressure to fractional inspired oxygen < 300
* Donor radiograph with 2 quadrant infiltrates
* Donor that are determined single lung donors prior to transplant will be excluded.

Recipient exclusion criteria

* Recipient age > 70 years.
* Recipient history of pulmonary hypertension (idiopathic pulmonary arterial hypertension, or secondary pulmonary arterial hypertension with mean arterial pressure > 30 mm Hg)
* Recipient history of abnormal cardiac function defined as prior coronary artery bypass graft (CABG) or left ventricular ejection fraction (LVEF) < 45 %
* Recipient history of open thoracotomy/prior pleurodesis as exclusion criteria. However patients who have had limited video-assisted thoracic surgery procedures for biopsies would NOT be excluded from the study.
* Recipient history of cirrhosis
* Recipient history of mechanical ventilation or extracorporeal support pre-operatively
* Recipient pre-operative hypotension defined by a systolic blood pressure less than 90 mm Hg not responsive to intravenous fluids or requirement for vasoactive medications
* Recipient preoperative history of renal insufficiency, dialysis or estimated glomerular filtration rate <30 ml/min/1.73 m2 body surface area
* Patients undergoing retransplantation
* Recipient history of significant coronary artery disease that is flow limiting and unable to be corrected by further percutaneous coronary artery interventions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Morrell, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Bobadilla JL, Love RB, Jankowska-Gan E, Xu Q, Haynes LD, Braun RK, Hayney MS, Munoz del Rio A, Meyer K, Greenspan DS, Torrealba J, Heidler KM, Cummings OW, Iwata T, Brand D, Presson R, Burlingham WJ, Wilkes DS. Th-17, monokines, collagen type V, and primary graft dysfunction in lung transplantation. Am J Respir Crit Care Med. 2008 Mar 15;177(6):660-8. doi: 10.1164/rccm.200612-1901OC. Epub 2008 Jan 3. PMID 18174545
- [Background] Christie JD, Van Raemdonck D, de Perrot M, Barr M, Keshavjee S, Arcasoy S, Orens J; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part I: introduction and methods. J Heart Lung Transplant. 2005 Oct;24(10):1451-3. doi: 10.1016/j.healun.2005.03.004. No abstract available. PMID 16210115
- [Background] Huang HJ, Yusen RD, Meyers BF, Walter MJ, Mohanakumar T, Patterson GA, Trulock EP, Hachem RR. Late primary graft dysfunction after lung transplantation and bronchiolitis obliterans syndrome. Am J Transplant. 2008 Nov;8(11):2454-62. doi: 10.1111/j.1600-6143.2008.02389.x. Epub 2008 Sep 10. PMID 18785961
- [Background] Kuntz CL, Hadjiliadis D, Ahya VN, Kotloff RM, Pochettino A, Lewis J, Christie JD. Risk factors for early primary graft dysfunction after lung transplantation: a registry study. Clin Transplant. 2009 Nov-Dec;23(6):819-30. doi: 10.1111/j.1399-0012.2008.00951.x. Epub 2009 Feb 20. PMID 19239481
- [Background] Prekker ME, Nath DS, Walker AR, Johnson AC, Hertz MI, Herrington CS, Radosevich DM, Dahlberg PS. Validation of the proposed International Society for Heart and Lung Transplantation grading system for primary graft dysfunction after lung transplantation. J Heart Lung Transplant. 2006 Apr;25(4):371-8. doi: 10.1016/j.healun.2005.11.436. Epub 2006 Feb 28. PMID 16563963
- [Background] Lee JC, Christie JD. Primary graft dysfunction. Proc Am Thorac Soc. 2009 Jan 15;6(1):39-46. doi: 10.1513/pats.200808-082GO. PMID 19131529
- [Background] Christie JD, Carby M, Bag R, Corris P, Hertz M, Weill D; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part II: definition. A consensus statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2005 Oct;24(10):1454-9. doi: 10.1016/j.healun.2004.11.049. Epub 2005 Jun 4. No abstract available. PMID 16210116
- [Background] de Perrot M, Bonser RS, Dark J, Kelly RF, McGiffin D, Menza R, Pajaro O, Schueler S, Verleden GM; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part III: donor-related risk factors and markers. J Heart Lung Transplant. 2005 Oct;24(10):1460-7. doi: 10.1016/j.healun.2005.02.017. Epub 2005 Aug 8. No abstract available. PMID 16210117
- [Background] Thabut G, Vinatier I, Stern JB, Leseche G, Loirat P, Fournier M, Mal H. Primary graft failure following lung transplantation: predictive factors of mortality. Chest. 2002 Jun;121(6):1876-82. doi: 10.1378/chest.121.6.1876. PMID 12065352
- [Background] Dejam A, Hunter CJ, Tremonti C, Pluta RM, Hon YY, Grimes G, Partovi K, Pelletier MM, Oldfield EH, Cannon RO 3rd, Schechter AN, Gladwin MT. Nitrite infusion in humans and nonhuman primates: endocrine effects, pharmacokinetics, and tolerance formation. Circulation. 2007 Oct 16;116(16):1821-31. doi: 10.1161/CIRCULATIONAHA.107.712133. Epub 2007 Sep 24. PMID 17893272

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Nitrite: Sodium Nitrite will be administered at three time points:
  At the time of organ procurement, a pre-prepared syringe of sodium nitrite will be added to each of the 2.8 Liter bags of Perfadex solution to flush the donor lungs.
  At the time of transplant just prior to reperfusion of lungs, , the donor lungs are flushed with a cold pneumoplegia solution after the bronchial (1st) anastomosis and with warm pneumoplegia solution after the portal vein (3rd, last) anastomosis. The drug will be added to pneumoplegia solution just prior to both the flushes.
  Sodium Nitrite will be delivered intravenously to the recipient immediately prior to lung reperfusion as a single infusion at rate of 4 mL/min for the first 30 min, followed by 2.2 mL/min for the next 60 min.
  Sodium Nitrite: Same as the details in Arm Description.
Period: Overall Study
Arm/Group | Sodium Nitrite
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety of Sodium Nitrite Administration Measured by Methemoglobin Levels
Description: The safety of Sodium Nitrite administration will be assessed by methemoglobin levels during and 150 minutes after the nitrite infusion in the transplant recipient.
Time Frame: 150 minutes post infusion
Measure: Mean (Standard Deviation); unit: percentage of methemoglobin
Groups:
- Sodium Nitrite: Sodium Nitrite will be administered at three time points:
  At the time of organ procurement, a pre-prepared syringe of sodium nitrite will be added to each of the 2.8L bags of Perfadex solution to flush the donor lungs.
  At the time of transplant just prior to reperfusion of lungs, , the donor lungs are flushed with a cold pneumoplegia solution after the bronchial (1st) anastomosis and with warm pneumoplegia solution after the PV (3rd, last) anastomosis. The drug will be added to pneumoplegia solution just prior to both the flushes.
  Sodium Nitrite will be delivered intravenously to the recipient immediately prior to lung reperfusion as a single infusion at rate of 4 mL/min for the first 30 min, followed by 2.2 mL/min for the next 60 min.
  Sodium Nitrite: Same as the details in Arm Description.
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
percentage of methemoglobin | 1.45 (0.35)

2. Primary Outcome: Safety of Sodium Nitrite Administration - Number of Participants With Fall in Patient's Mean Arterial Pressure Greater Than 20%
Description: The safety of Sodium Nitrite administration will be assessed by the incidence of fall in patient's Mean Arterial Pressure greater than 20% from recorded baseline requiring discontinuation of drug infusion during and after the nitrite infusion in the transplant recipient. Mean Arterial Pressure will be monitored at 1 minute intervals during study drug infusion followed by 15 minute intervals for 1 hour.
Time Frame: Baseline and 1 hour post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Number of Participants With Primary Graft Dysfunction Grades 2+3
Description: The primary study endpoint is the incidence of grades 2+3 Primary Graft Dysfunction (PGD) based upon the worst PGD grade during the first 72 hours post organ reperfusion. The severity of PGD is graded 0-3 based on the presence or absence of diffuse opacities on chest radiograph and the ratio of arterial oxygen pressure to inspired oxygen concentration. The grading system predicts post-lung transplant outcomes with Grade 3 being the worst.
Time Frame: First 72 hours post organ reperfusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Number of Participants With Acute Rejection
Description: To evaluate the efficacy of Sodium Nitrite infusion into the procured lungs and the lung transplant recipient in the prevention of delayed allograft complications including the incidence of acute rejection. Prevention of delayed allograft complications include clinically indicated spirometric and lung volume assessments of lung function performed as an indicator of Bronchiolitis Obliterans Syndrome (BOS), and evidence of pathological rejection by surveillance transbronchial lung biopsies.
Time Frame: Up to 12 months post lung transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
Participants | 1

5. Secondary Outcome: Number of Participants With Chronic Rejection
Description: To evaluate the efficacy of Sodium Nitrite infusion into the procured lungs and the lung transplant recipient in the prevention of delayed allograft complications including the incidence of chronic rejection. Prevention of delayed allograft complications include clinically indicated spirometric and lung volume assessments of lung function performed as an indicator of Bronchiolitis Obliterans Syndrome (BOS), and evidence of pathological rejection by surveillance transbronchial lung biopsies.
Time Frame: Up to 12 months post lung transplant
Measure: Count of Participants; unit: Participants
Groups:
- Sodium Nitrite: Sodium Nitrite will be administered at three time points:
  At the time of organ procurement, a pre-prepared syringe of sodium nitrite will be added to each of the 2.8L bags of Perfadex solution to flush the donor lungs.
  At the time of transplant just prior to reperfusion of lungs, the donor lungs are flushed with a cold pneumoplegia solution after the bronchial (1st) anastomosis and with warm pneumoplegia solution after the PV (3rd, last) anastomosis. The drug will be added to pneumoplegia solution just prior to both the flushes.
  Sodium Nitrite will be delivered intravenously to the recipient immediately prior to lung reperfusion as a single infusion at rate of 4 mL/min for the first 30 min, followed by 2.2 mL/min for the next 60 min.
  Sodium Nitrite: Same as the details in Arm Description.
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Number of Ventilator Free Days (VFD)
Description: Defined as the number of days off mechanical ventilation at baseline through Day 30 post transplantation.
Time Frame: Baseline through Day 30 post transplantation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
days | 18 (15.6)

7. Secondary Outcome: Number of ICU Free Days (IFD)
Description: Defined as the number of days outside the ICU through Day 30 post transplantation.
Time Frame: Day 30 post transplantation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 3
days | 14.7 (13.3)

ADVERSE EVENTS:
Time Frame: From study enrollment to 72 hours after the last dose of study drug, an average of 1 year
Arm/Group | Sodium Nitrite
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Nitrite (N=3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Nitrite (N=3)
Atypical appearance of the lungs (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early due to lack of funding support, difficulty in recruiting patients and lack of support staff. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT01715883/Prot_SAP_000.pdf